CLINICAL TRIAL: NCT01100723
Title: Trial to Optimize Mineral Outcomes in End Stage Renal Disease (ESRD) Patients
Brief Title: Trial to Optimize Mineral Outcomes in Dialysis Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 09-0623
Record Dates: First submitted 2010-04-07; First posted 2010-04-09 (Estimated); Results first posted 2017-01-02 (Estimated); Last update posted 2017-01-02 (Estimated); Status verified 2016-11

CONDITIONS: Secondary Hyperparathyroidism; Chronic Kidney Disease
Keywords: secondary hyperparathyroidism; calcium; phosphorus; ESRD; CKD; mineral disorder
MeSH Terms: conditions — Hyperparathyroidism, Secondary; Renal Insufficiency, Chronic; Kidney Failure, Chronic | interventions — Cinacalcet; paricalcitol; 1 alpha-hydroxyergocalciferol; Calcitriol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Computer directed dosing decisions (Experimental): This study will be an open-label, non-randomized, single arm design. Patients will have their mineral and bone disorders managed by the computer directed algorithm. The computer algorithm will make recommendations for dosing active vitamin D and cinacalcet. The doses of these medications recommended by the algorithm will then be prescribed to the subjects participating in the study unless overridden by the patients primary attending nephrology for other clinical or safety concerns. At any time in the study, subjects may be on neither, one, or both of these medication depending on their laboratory results and the output recommendations of the algorithm.
  Interventions: Other: Cinacalcet, active vitamin D analogue

INTERVENTIONS:
Other: Cinacalcet, active vitamin D analogue — Patients will have their mineral and bone disorders managed by the computer directed algorithm. Cinacalcet will be dose increased starting at 30 mg/day as indicated by protocol along with active vitamin D based on values of serum calcium, phosphorus and parathyroid hormone.
  Other Names: sensipar, paricalcitol, doxercalciferol, calcitriol

SUMMARY:
This trial is designed to determine if the use of a computer algorithm designed to optimize mineral outcomes in dialysis patients increases the number of patients achieving the desired target endpoints for calcium, phosphorus and parathyroid hormone.

DETAILED DESCRIPTION:
It is our hypothesis that a computerized dosing protocol incorporating both cinacalcet and vitamin D analogues can achieve significantly better control of mineral and bone parameters than currently observed in most dialysis facilities. This trial will test this hypothesis.

Objectives Primary Objectives

1. Compare the percent of patients achieving an intact parathyroid hormone (PTH) target of ≤ 300 pg/ml before and after the application of a computerized dosing protocol for management of chronic kidney diseases mineral and bone disorder (CKD-MBD).
2. Compare the percent of patients achieving a phosphorus of ≤ 5.5 mg/dL before and after the application of a computerized dosing protocol for management of CKD-MBD.

Secondary Objectives

1. Compare the percent of patients achieving an intact PTH target of ≤ 450 pg/ml before and after the application of a computerized dosing protocol for management of CKD-MBD.
2. Compare the percent of patients achieving a phosphorus of ≤ 4.5 mg/dL before and after the application of a computerized dosing protocol for management of CKD-MBD.
3. Compare the percent of patients achieving a calcium ≤ 10.1 mg/dL before and after the application of a computerized dosing protocol for management of CKD-MBD.
4. Compare the percent of patients on cinacalcet and vitamin D analogues at baseline and at 6 and 12 months after the application of a computerized dosing protocol for management of CKD-MBD.
5. Compare the mean and standard deviation (SD) at baseline and 6 and 12 months for PTH, calcium and phosphorus.
6. Compare the total monthly and average weekly (for patients on the medication) active vitamin D analogue dose at baseline and at 6 and 12 months (converted to mcg per month of paricalcitol) after the application of a computerized dosing protocol for management of CKD-MBD. 1 mcg paricalcitol = 0.5 mcg doxercalciferol
7. Compare the number of patients on calcium and non-calcium binders at baseline and at 6 and 12 months after the application of a computerized dosing protocol for management of CKD-MBD.
8. Determine the percent of patients who are non-compliant with oral cinacalcet and the percent that are unable to tolerate the dose required by the algorithm to achieve target outcomes

ELIGIBILITY:
Inclusion Criteria:

* Men or women 18 years of age or older
* On outpatient hemodialysis
* Have a level of understanding and willingness to cooperate with the study personnel
* Able to provide informed consent

Exclusion Criteria:

* Currently enrolled in another interventional clinical trial
* Are pregnant, plan on becoming pregnant during the study period, or breast-feeding
* Planned parathyroidectomy within 6 months
* Planned kidney transplant within 6 months
* Life expectancy < 6 months
* Patient declines participation
* Liver function tests > 2 times the upper limit of normal

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2010-03; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David M Spiegel, MD, Principal Investigator — University of Colorado, Denver
Locations (1):
- Lynchburg Nephrology Associates, P.L.L.C., Lynchburg, Virginia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Spiegel DM, McPhatter L, Allison A, Drumheller JC, Lockridge R. A computerized treatment algorithm trial to optimize mineral metabolism in ESRD. Clin J Am Soc Nephrol. 2012 Apr;7(4):632-9. doi: 10.2215/CJN.08170811. Epub 2012 Feb 2. PMID 22300740

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 181 pts in dialysis center. 65 did not meet enrollment criteria. 23 declined participation and 1 had prior intolerance to cinacalcet. Therefore 92 subjects enrolled in study.
Pre-assignment Details: No washout. Once enrolled, mineral and bone disorder managed by computer algorithm.
Groups:
- Post Treatment: Patients had their mineral and bone disorders managed by the computer directed algorithm. Cinacalcet dose was increased starting at 30 mg/day as indicated by protocol along with active vitamin D based on values of serum calcium, phosphorus and parathyroid hormone.
Period: Overall Study
Arm/Group | Post Treatment
Started | 92
6 Month Analysis | 85 (85 subjects had laboratory data at the 6 month analysis and were compared to their baseline data.)
Completed | 78 (78 subjects had laboratory data at the 12 month analysis and were compared to their baseline data.)
Not Completed | 14

BASELINE CHARACTERISTICS:
Groups:
- Post Treatment: Results analyzed at study evaluation time points.
Arm/Group | Post Treatment
Number analyzed (Participants) | 92
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 60
  >=65 years | 32
Gender [Count of Participants; unit: Participants]
  Female | 40
  Male | 52

OUTCOME MEASURES:

1. Primary Outcome: Percent of Patients Achieving Parathyroid Hormone Target ≤ 300
Description: Compare the percent of patients achieving an intact Parathyroid hormone (PTH) target of ≤ 300 pg/ml before and after the application of a computerized dosing protocol for management of chronic kidney disease-mineral and bone disorder (CKD-MBD). If multiple values were obtained within a specified evaluation time frame the values were averaged and the average value was then evaluated as to whether it was within or outside the target range.
Time Frame: 1 year
Population: Subjects who had at least one laboratory measurement during the assessment phase.
Measure: Number; unit: percentage of subjects meeting target
Arm/Group | Post Treatment
Number analyzed (Participants) | 78
percentage of subjects meeting target | 21
Statistical Analysis 1: Comparison: Post Treatment; Number of subjects meeting targets were compared to the same subjects baseline values using the McNemar test for paired longitudinal data. For the 1 year analysis, the proportion of subjects with PTH values in the target range was calculated at 1 year and that was compared to the proportion of the same subjects who were in target at baseline; Test type: Superiority or Other; p < 0.05, McNemar

2. Primary Outcome: Percent of Patients Achieving Phosphorous Target ≤ 5.5
Description: Compare the percent of patients achieving a phosphorus of ≤ 5.5 mg/dL before and after the application of a computerized dosing protocol for management of CKD-MBD. If multiple values were obtained within a specified evaluation time frame the values were averaged and the average value was then evaluated as to whether it was within or outside the target range.
Time Frame: 1 year
Measure: Number; unit: percent of participants in target
Groups:
- Results Analyzed at Study Evaluation Time Points.: Results analyzed at study evaluation time points of 1 year and 6 months.
Arm/Group | Results Analyzed at Study Evaluation Time Points.
Number analyzed (Participants) | 78
percent of participants in target | 53
Statistical Analysis 1: Comparison: Results Analyzed at Study Evaluation Time Points; Number of subjects meeting targets were compared to the same subjects baseline values using the McNemar test for paired longitudinal data. For the 1 year analysis, the proportion of subjects with phosphorus values in the target range was calculated at 1 year and that was compared to the proportion of the same subjects who were in target at baseline; Test type: Superiority or Other; p < 0.05, McNemar

3. Secondary Outcome: Percent of Patients Achieving Parathyroid Hormone Target ≤ 450
Description: Compare the percent of patients achieving an intact PTH target of ≤ 450 pg/ml before and after the application of a computerized dosing protocol for management of CKD-MBD. If multiple values were obtained within a specified evaluation time frame the values were averaged and the average value was then evaluated as to whether it was within or outside the target range.
Time Frame: 1 year
Measure: Number; unit: percent of participants in target
Arm/Group | Post Treatment
Number analyzed (Participants) | 78
percent of participants in target | 33
Statistical Analysis 1: Comparison: Post Treatment; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.05, McNemar

4. Secondary Outcome: Percent of Patients Achieving Phosphorous Target ≤ 4.5
Description: Compare the percent of patients achieving a phosphorus of ≤ 4.5 mg/dL before and after the application of a computerized dosing protocol for management of CKD-MBD. If multiple values were obtained within a specified evaluation time frame the values were averaged and the average value was then evaluated as to whether it was within or outside the target range.
Time Frame: 1 year
Measure: Number; unit: percent of participants in target
Arm/Group | Post Treatment
Number analyzed (Participants) | 78
percent of participants in target | 29
Statistical Analysis 1: Comparison: Post Treatment; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p < 0.05, McNemar

5. Secondary Outcome: Percent of Patients Achieving Calcium Target ≤ 10.1
Description: Compare the percent of patients achieving a calcium ≤ 10.1 mg/dL before and after the application of a computerized dosing protocol for management of CKD-MBD. If multiple values were obtained within a specified evaluation time frame the values were averaged and the average value was then evaluated as to whether it was within or outside the target range.
Time Frame: 1 year
Population: Subjects with at least one laboratory value during evaluation period.
Measure: Number; unit: percentage of subjects in target
Arm/Group | Post Treatment
Number analyzed (Participants) | 78
percentage of subjects in target | 78
Statistical Analysis 1: Comparison: Post Treatment; Number of subjects meeting targets were compared to the same subjects baseline values using the McNemar test for paired longitudinal data. For the 1 year analysis, the proportion of subjects with Ca values in the target range was calculated at 1 year and that was compared to the proportion of the same subjects who were in target at baseline; Test type: Superiority or Other; p < 0.05, McNemar

6. Secondary Outcome: Percent of Patients on Cinacalcet and Vitamin D Analogues
Description: Compare the percent of patients on cinacalcet and vitamin D analogues at baseline and at 6 and 12 months after the application of a computerized dosing protocol for management of CKD-MBD. If multiple values were obtained within a specified evaluation time frame the values were averaged and the average value was then evaluated as to whether it was within or outside the target range.
Time Frame: 6 months and 1 year
Population: Number of subjects with at least 1 laboratory analysis during the evaluation period.
Measure: Number; unit: percentage of subjects receiving med
Arm/Group | Post Treatment
Number analyzed (Participants) | 78
percentage of subjects receiving med | 84
Statistical Analysis 1: Comparison: Post Treatment; Proportion of subjects on specified medications were compared to the same subjects baseline values using the McNemar test for paired longitudinal data. For the 1 year analysis, the proportion of subjects on the specified medications was calculated at 1 year and that was compared to the proportion of the same subjects who were in target at baseline; Test type: Superiority or Other; p < 0.05, McNemar

ADVERSE EVENTS:
Arm/Group | Post Treatment
Serious Adverse Events (participants affected / at risk) | 0/92
Other Adverse Events (participants affected / at risk) | 0/92

LIMITATIONS AND CAVEATS:
No adverse events reported. Dose titration limited by hypocalcemia and subject non-adherent to oral medications.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No